CLINICAL TRIAL: NCT06307509
Title: Changes in Adipose Tissue Structure and Function in the Context of Sepsis
Brief Title: Adiposity and Immunometabolism in Sepsis
Acronym: AIMS
Status: Not yet recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN23AN097
Record Dates: First submitted 2024-02-13; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Obesity; Sepsis
Keywords: obesity; adipose tissue; sepsis; critical illness
MeSH Terms: conditions — Obesity; Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen subcutaneous and visceral adipose tissue samples, isolated adipocytes and serum samples will be retained and stored as per University of Glasgow protocols
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU patients with sepsis: Patients admitted to the Intensive Care Unit with a primary diagnosis of sepsis. They will have subcutaneous adipose tissue samples taken by needle aspiration, and blood samples taken.
  Interventions: Other: Diagnosis of sepsis
- Surgical patients with sepsis: Patients undergoing emergency laparotomy with a diagnosis of sepsis will have subcutaneous and visceral adipose tissue samples taken intra-operatively, and blood samples taken.
  Interventions: Other: Diagnosis of sepsis

INTERVENTIONS:
Other: Diagnosis of sepsis — Patients will be recruited on the basis of a diagnosis of sepsis, as this is the exposure of interest

SUMMARY:
Obesity has been shown to increase adverse outcomes in some critically ill patients e.g. those with COVID-19. For patients with sepsis this association is less clear cut but there is evidence that body fat distribution, resulting from impaired subcutaneous adipose tissue function, is associated with adverse clinical outcomes in critical care. The investigators aim to study subcutaneous adipose tissue function in lean and obese sepsis patients in critical care and compare that to healthy controls.

First, the study will investigate differences in adipose tissue function (inflammation and mitochondrial function) related to obesity. Second, the investigators will examine whether lean critically ill patients with sepsis have enhanced adipose tissue inflammation and mitochondrial dysfunction compared to lean controls and whether this is further exacerbated by obesity.

Patients will be either undergoing emergency abdominal surgery, or will have been admitted to a critical care unit with a diagnosis of sepsis.

The investigators will collect blood and adipose tissue biopsies from the patients, and these will be analysed for markers of inflammation and of mitochondrial function.

The aim is to better understand the relationship between obesity, inflammation, mitochondrial dysfunction and sepsis. The investigators hope that this may improve the understanding of the pathophysiology of sepsis and allow more targeted interventions for patients based on differences in their baseline metabolic state.

DETAILED DESCRIPTION:
Hypothesis The hypothesis is that adipose tissue from patients who are critically ill with sepsis will show changes in structure, increased inflammatory function, and increased mitochondrial dysfunction in comparison to control patients without sepsis. The investigators also hypothesise that that increased inflammatory function will be more pronounced in VAT than in SAT.

Aims The investigators aim to investigate potential differences in adipose tissue structure, inflammatory function, and mitochondrial dysfunction between individuals with and without sepsis, and between SAT and VAT.

Study design

There will be two patient cohorts:

1. Patients undergoing emergency surgery with a diagnosis of sepsis

   a. 15-30 patients
2. Patients admitted to a critical care unit with a diagnosis of sepsis

   1. 15-30 patients

      Results from patients with sepsis will be compared with results obtained from a cohort of patients recruited to a previous study (CONNECT study: IRAS project ID 291251; REC reference 21/NS/0015). These patients are recruited when undergoing an elective abdominal operation, with no evidence of an acute inflammatory process. When recruited to the study, they undergo an identical fat and blood sampling process to that described in this study.

      Study Setting Patients will be recruited from the operating theatre suite and the Critical Care Units at the Queen Elizabeth University Hospital Glasgow.

      Adipose tissue samples will only be taken from those who require sedation or general anaesthesia for tracheal intubation, either in the critical care unit, or in the operating theatre.

      Consent Consent process Patients in ICU, particularly in the acute phase of their illness, often lack decision-making capacity due to delirium and the effects of sedative medications. In order to evaluate the changes that take place in adipose tissue during the acute phase of critical illness, it is important to undertake sampling as soon as possible after a patient's admission to an ICU. It is anticipated that the patients recruited in ICU in this study will not be able to consent prospectively to enrolment in this study. Therefore, a researcher will seek consent from a Welfare Attorney, Welfare Guardian or nearest relative. This researcher will be trained in consent procedures that adhere to the ethical principles in the Declaration of Helsinki and the Adults with Incapacity Act (2000) Scotland. The researcher will provide the study Information Sheet, and the Consent Form, and will review the contents to ensure that the procedures, benefits, and risks of the study are understood. The person being approached will be asked to give their consent based on their perception of the wishes of the patient if they had capacity. They will then be invited to sign the consent form. The original will be retained in the investigator site file, and a copy given to the person who signed the form and another copy placed in the patients' medical records.

      Patient consent to continue Patients consented to the study by a Welfare Attorney, Welfare Guardian or nearest relative will be approached to obtain their permission to continue in the study once they have recovered capacity after their critical illness. Patients will be approached by an appropriately trained member of the research team, and provided with the study Information Sheet, and a copy of the Consent to Continue form. The researcher will review the contents of these with the patient, provide clarification and an opportunity for questions. Patients who decline to participate at this stage will be removed from the study.

      Withdrawal from the study Participants may withdraw from the study at any point without suffering any disadvantage.

      Study procedures Clinical data collection

      Baseline data will be collected for all patients recruited to the study. This will include, but is not limited to:
      * Age
      * Sex
      * BMI
      * Major comorbidities

      For patients admitted to an ICU, further data will be collected with regards to their acute illness. This will include, but is not limited to:
      * APACHE II
      * Biochemical & haematological parameters, where measured clinically:

        * Highest C-reactive protein in first 48 hours
        * Highest white cell count in first 48 hours
        * Highest procalcitonin in first 48 hours
        * Highest lactate in first 48 hours
      * Physiological parameters:

        * Highest heart rate in first 48 hours (in beats per minute)
        * Highest noradrenaline dose in first 48 hours (in mcg/min)
        * Lowest P:F ratio in first 48 hours
        * Highest dose of insulin delivered in first 48 hours (in units/hr)
      * Outcome data:

        * ICU length-of-stay
        * ICU outcome
        * Number of days requiring invasive mechanical ventilation
        * Number of days requiring cardiovascular support
        * Number of days requiring renal replacement therapy
        * Hospital length-of stay
        * Hospital outcome

      Imaging data collection

      The investigators will review the clinical imaging acquired for each patient recruited into the study. Any patient who has undergone a CT scan, which includes the L3 vertebral level, in the 12 months preceding their admission to an ICU, or the 48 hours following their admission, will be suitable for CT-derived body composition analysis. A single image slice at the level of the L3 vertebra will be obtained. This image will then be deidentified and downloaded from PACS to an NHS Greater Glasgow and Clyde computer. The deidentified image will then be uploaded to the CoreSlicer software programme, and analysed as described previously (35). This will allow calculation of the area of visceral adipose tissue, subcutaneous adipose tissue, and muscle mass. This may provide a more nuanced assessment of an individual's adiposity than BMI alone.

      Blood and adipose tissue sampling Blood Sampling Up to 40ml of blood will be collected by trained staff at recruitment to the study.

      Adipose tissue sampling in patients in a critical care unit Adipose tissue will be taken 5 cm lateral to the umbilicus under sterile conditions using a 20ml Terumo™ Luer Tip Syringe attached to a 14G 80mm Sterican Single Use Deep Intramuscular Needle prefilled with approximately 5ml of 0.9% saline. Each biopsy pass collects on average 0.3g tissue, so three passes should provide up to 1g adipose tissue. This will be filtered through a 100μm nylon mesh filter and transported to the laboratory in 15ml of pre-warmed (370C) Gibco™ Medium 199, Hanks' Balanced Salts solution.

      Adipose tissue sampling in patients undergoing emergency surgery Both subcutaneous and visceral adipose tissue will be taken under direct vision by the surgical team. Approximately 1g of tissue will be taken by from each site. This will be transported to the laboratory in 15ml of pre-warmed (370C) Gibco™ Medium 199, Hanks' Balanced Salts solution.

      Transportation of samples to the University of Glasgow All samples (blood and adipose tissue) will be packaged for transport to the University of Glasgow in accordance with the current Health Protection Scotland guidance.

      Expected duration of subject participation The whole procedure, including blood sampling and adipose sampling, should take less than 30 minutes.

      Adipose tissue analysis From a 1g adipose tissue biopsy, 300µl 90% cytocrit adipocytes and a stromovascular fraction (SVF) can be prepared. If additional adipose tissue is available, this will be flash frozen in liquid nitrogen and stored at -800C for later histological analysis.

      Adipocyte sizing will be carried out on unfixed fresh adipocyte suspensions (5µL) isolated by collagenase digestion of the biopsy, imaged on an Olympus BX50 microscope using a x10 lens connected to 3-CCD colour camera (JVC) for digital image capture with Image J automated sizing.

      Basal and lipopolysaccharide (1µM) stimulated adipokine secretion, corrected for cell number using adipocyte suspension DNA concentrations (isolated concurrently with RNA), will be assessed in isolated adipocytes (in duplicate 50µL per assay) after 2 hours at 37°C, as described previously (36).

      Adipocyte inflammatory gene expression will be quantitated relative to the endogenous control PPIA in RNA isolated from adipocyte suspension (95µL, yielding approximately 500ng RNA) using TRIzol (ThermoFisher Scientific). Chosen targets will be pre-amplified in the RNA followed by Taqman RT-PCR quantitation using commercial primer probes sets (ThermoFisher Scientific).

      SVF cells will be cultured in 25 cm2 flasks, in a 37°C 5% CO2 incubator, in Dulbecco's Modified Eagle Medium (DMEM) and sampled at 2 and 24 hours for analysis of cytokines. The culture (passage 0) will be continued to allow pre-adipocytes to adhere, changing medium every 3-4 days until 80% confluent when the preadipocyte will be passaged until 80% confluent (passage 1). At the end of passage 1 pre-adipocytes will be detached and frozen at 500,000 cells/mL in DMEM, 20% FBS, 10% dimethyl sulfoxide [DMSO, DLM-10RG-PK], 100 U/mL penicillin-streptomycin, and 2 mM L-Glutamine) and stored in liquid nitrogen for later analysis of pre-adipocyte differentiation.

      Cytokine quantitation will be carried out using magnetic bead multiple arrays (Merck Millipore) on a MAGPIX® xPONENT 4.2 system or by commercial ELISA.

      Adipose tissue vascularisation and fibrosis will be assessed on available frozen biopsies embedded in OCT. Cryosections (10µm) will be immunostained using anti-CD31 to identify blood vessels. Blood vessel density will be calculated as the ratio of blood vessel number to total section area. Adipose tissue fibrosis will be assessed using picosirius red and Image J analysis.

      Adipocytes will be stained with MitoTracker Green FM and MitoTracker Red, according to manufacturer's instructions, and imaged using fluorescence microscopy in the BHF GCRC Imaging Suite. Images will be analysed to assess mitochondrial morphology (interconnectivity, size and swelling) using Mitomorph software. Adipocyte mitochondria content will also be assessed after JC-1 staining as fluorescence intensity per cell in a Cellometer. Mitochondrial content will be confirmed using the independent method of mtDNA/nuclear DNA ratio using MT-CO2, MT-CYB, PPARG and UCP1 expression by Taqman RT-PCR.

      Mitochondrial fission/fusion will be estimated by quantifying the expressions of genes/proteins involved in mitochondrial fission (DNM1L) and fusion (MFN1, MFN2 and RHOT1) using Taqman RT-PCR and western blotting.

      Gene and protein expression of mitochondrial respiratory complex and fatty acid oxidation proteins will be carried out using Taqman RT-PCR and western blotting respectively.

      Blood sample analysis Plasma will be separated and frozen in aliquots at -80 degrees Celsius. Plasma adipokine (e.g. adiponectin, visfatin) levels will be measured using commercial ELISA, as per standard product protocols.

      Clinical management of patients in the study There will be no changes to patients' clinical management as part of this study.

      Assessment of safety Definitions of Adverse Events Adverse Events (AEs) and Serious Adverse Events (SAEs) are defined as per the International Conference on Harmonisation Good Clinical Practice (ICH-GCP) glossary of terms.

      Adverse Events Needle punctures for blood and adipose tissue sampling do not cause any serious problems for most patients. There is a small risk that needle punctures may cause dizziness, discomfort, bleeding, bruising, or infections at the site.

      Recording and reporting of Adverse Events Any untoward medical occurrence in a patient involved in the study related to sample collection will be recorded and reported in accordance with the Research Governance Framework (i.e. annually for AEs and within 15 days for SAEs). Any SAE which is unexpected and related to the sample collection will be reported to the Research Ethics Committee within 15 days of the Chief Investigator becoming aware of the event. A summary of AEs and SAEs will be provided to the Research Ethics Committee and the Research & Development Office, NHS GGC, annually. The AEs and SAEs will be collected in the case report forms during the period of the study.

      Data Collection & Management Direct access to source data/documents Patient specific information will be accessed from the electronic patient data management system (IntelliSpace Critical Care and Anesthesia, Phillips Medical Systems) and from the Clinical Portal electronic patient record. Access to these data systems for the purpose of the study will be limited to appropriately delegated members of the study team. Access by internal or external auditors will be managed in accordance with the relevant Standard Operating Procedures of the Glasgow Clinical Research Facility.

      Data centre All identifiable data collected within the NHS Greater Glasgow and Clyde (NHS GGC) will remain within NHS GGC. Only anonymised data and tissue samples will be shared with the University of Glasgow.

      All tissue samples will be processed and analysed at the University of Glasgow School of Cardiovascular and Metabolic Health (SCMH), and surplus samples bio-banked. The bio-banked tissue samples and associated data will be stored and used in accordance with the policies of the SCMH.

      Data Access Requests to access the data generated in this study should be made to the Chief Investigator, and will be considered on an individual case-by-case basis, and will be discussed with the Sponsor.

      Data Retention Data will be retained for 5 years following completion of the study and will remain the responsibility of the Chief Investigator.

      Quality assurance During and/or after completion of the study, quality assurance officers named by NHS GGC or the regulatory authorities may wish to perform onsite audits. The Principal Investigator will be expected to cooperate with any audit and to provide assistance and documentation (including source data) as requested.

      Statistics Sample size A total of 60 patients will be recruited, with 30 patients undergoing emergency surgery, and 30 patients who have been admitted to a critical care unit. (as detailed under Study design above).

      The inflammatory function of adipose tissue has not been examined in human tissue in patients with sepsis in critical care. Previous work found significant differences in adipocyte insulin resistance, adipokine secretion and genes expression between pre-eclampsia patients and healthy pregnancy with n=13 patients per group (36,37). Unpublished data comparing subcutaneous adipocyte differentiation between age and BMI-matched European and South Asian men found an PPARγ effect size of 0.72 (calculated using GPower). Assuming the study might find a similar effect size between sepsis patients and controls, the investigators require n=25 participants to detect a similar level of difference in gene expression with 80% power. Accordingly, the investigators anticipate n=30 patients per group will be sufficient to show significant differences in adipocyte function for the proposed study, allowing for some incomplete analyses.

      Description of statistical methods The primary outcome will be analysed using a 2-way ANOVA mixed model. Independent variables will be the presence or absence of sepsis, and the adipose tissue depot sampled (subcutaneous and visceral). The dependent variable will be quantity of cytokine secreted. The investigators will include covariates in the model that are known to influence adipose tissue distribution and function such as age, gender, BMI and, where available, ratio of SAT:VAT (as a measurement of adipose tissue distribution).

      For analyses in which both SAT and VAT are not available, populations will be compared using two-sample t-tests where data is normally distributed (or can be transformed to achieve this) or the Mann Whitney u-test if non-parametrically distributed.

      Level of significance to be used A p-value of <0.05 will be considered statistically significant. All secondary analyses will be purely exploratory and should be interpreted as hypothesis-generating.

      Ethics & Clinical Governance Ethical approval This protocol and any amendments will be submitted to the Scotland A Research Ethics Committee (REC), with the authority to review studies requiring approval under the Adults with Incapacity (Scotland) Act 2000. A copy of the documented decision of the REC will be available to the sponsor and appropriate Research & Development (R&D) offices at each of the sites for their formal approval of the study. Only sites which have been granted ethics approval through the site-specific assessment, and R&D management approval will be allowed to initiate the study.

      Statement of compliance This study will adhere to the principles of the Data Protection Act and the General Data Protection Regulations (GDPR), The Declaration of Helsinki, and all relevant guidelines and legislation governing clinical research. The investigators are responsible for the conduct of the study in accordance with the principles of the International Conference on Harmonisation Good Clinical Practice (ICH-GCP) guidelines (www.ich.org). All members of the study team will be required to have completed GCP training.

      Informed consent The vulnerability of this study group is fully appreciated, and every effort will be undertaken to protect their safety and well-being. In line with the applicable regulatory requirements and to comply with the Research Governance Framework, consenting processes will be standardised and a robust Standard Operating Procedure for consenting patients will be adhered to. The first contact will be by clinical staff caring for the patient.

      Patient confidentiality To maintain confidentiality, all case report forms (CRFs), study reports and communication regarding the study will identify the patients by the assigned unique study identifier and initials only. Patient confidentiality will be maintained at every stage and data will not be made publicly available to the extent permitted by the applicable laws and regulations.

      Sponsorship This study will be sponsored by NHS Greater Glasgow & Clyde Research & Innovation.

ELIGIBILITY:
Inclusion Criteria:

For patients in a critical care unit:

Diagnosis of sepsis by the criteria set out in the Sepsis-3 guidelines:

1. Suspected diagnosis of infection
2. Acute change in Sequential Organ Failure Assessment (SOFA) of ≥2

For patients undergoing an operation:

Undergoing emergency abdominal surgery

Diagnosis of sepsis by the criteria set out in the Sepsis-3 guidelines:

1. Suspected diagnosis of infection
2. Acute change in Sequential Organ Failure Assessment (SOFA) of ≥2

Exclusion Criteria:

* Patient moribund and death is perceived to be imminent
* ≥48 hours from diagnosis with sepsis
* Pregnancy
* Prisoners
* Receiving treatment-dose anticoagulant medication
* Declined consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a critical care unit with a diagnosis of sepsis will be screened using the IntelliSpace Critical Care and Anesthesia electronic patient record, after identification and discussion with the clinical team.
  Patients undergoing emergency surgery will be screened using the Opera theatre management system, after identification and discussion with the clinical teams.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Difference in adipocyte cytokine secretion between patients with sepsis, and patients without sepsis, and between SAT and VAT samples | Within 72 hours of admission to ICU
  Cytokine quantitation from adipose tissue samples will be carried out using using magnetic bead multiple arrays or by commercial ELISA to investigate for any possible differences between patients with and without sepsis, and between SAT and VAT samples

SECONDARY OUTCOMES:
Differences in adipocyte size | Within 72 hours of admission to ICU
  Between patients with and without sepsis, and between SAT and VAT samples
Differences in mitochondrial morphology | Within 72 hours of admission to ICU
  Between patients with and without sepsis, and between SAT and VAT samples
Differences in adipocyte pro-inflammatory gene expression | Within 72 hours of admission to ICU
  Between patients with and without sepsis, and between SAT and VAT samples
Differences in adipocyte mitochondrial number | Within 72 hours of admission to ICU
  Between patients with and without sepsis, and between SAT and VAT samples
Differences in adipocyte mitochondrial viability | Within 72 hours of admission to ICU
  Between patients with and without sepsis, and between SAT and VAT samples
Differences in SVF cytokine secretion | Within 72 hours of admission to ICU
  Between patients with and without sepsis, and between SAT and VAT samples
Differences in capacity of pre-adipocytes to differentiate into mature adipocytes | Within 72 hours of admission to ICU
  Between patients with and without sepsis, and between SAT and VAT samples

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Watson, MBChB, PhD, Principal Investigator — NHS Greater Glasgow & Clyde
Locations (1):
- Department of Critical Care Medicine, Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No